CLINICAL TRIAL: NCT02836509
Title: Comparison of Intravenous Ibuprofen and Paracetamol in Patients With Low Back Pain Presented to the Emergency Department: A Randomized, Double-Blind, Controlled Trial
Brief Title: Comparison of Intravenous Ibuprofen and Paracetamol in Patients With Low Back Pain Presented to the Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Mustafa Serinken, professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: LBPainIvsP
Record Dates: First submitted 2016-07-01; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Ibuprofen; Paracetamol; Emergency Medicine
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paracetamol group (Experimental): First Group: 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes. (100 ml of saline is removed before the addition of the 100 ml paracetamol to be the same volume)
  Interventions: Drug: Paracetamol
- Ibuprofen group (Experimental): Second Group: 800 mg Ibuprofen in 150 ml normal saline given as a slow intravenous infusion over 5 minutes
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes.
  Other Names: PERFALGAN; PARTEMOL; PAROL
  Arms: paracetamol group
Drug: Ibuprofen — 800 mg Ibuprofen in 150 ml normal saline given as a slow intravenous infusion over 5 minutes
  Other Names: intrafen; Caldolon
  Arms: Ibuprofen group

SUMMARY:
Currently, Paracetamol and Ibuprofen are widely used by emergency physicians in Turkey for the pain treatments.

The objective of the study was to assess whether intravenous Paracetamol has superior Low Back Pain reduction will compare with Ibuprofen in emergency department (ED) adults.

Half of the participants will receive Paracetamol and the other half will receive Ibuprofen.

DETAILED DESCRIPTION:
Paracetamol and Ibuprofen each relieve pain with different mechanisms.

Paracetamol is termed a simple analgesic and an antipyretic. Despite enduring assertions that it acts by inhibition of cyclooxygenase (COX)-mediated production of prostaglandins, unlike non-steroidal anti-inflammatory drugs (NSAIDs).

Ibuprofen is the most commonly used and most frequently prescribed NSAID. It is a non-selective inhibitor of cyclo-oxygenase-1 (COX-1) and Cyclooxygenase-2 (COX-2).4 Although its anti inflammatory properties may be weaker than those of some other NSAIDs, it has a prominent analgesic and antipyretic role.

In the investigators trial; The investigators aimed to compare intravenous Paracetamol and Ibuprofen in patient with Low Back Pain

* All patients eligible for the study were randomized to one of two groups:
* First Group: 1000 mg Paracetamol in 150 ml normal saline given as a slow intravenous infusion over 5 minutes.
* 100 ml of saline is removed before the addition of the 100 ml paracetamol (Perfalgan, Bristol Myers, Italy) to be the same volume.
* Second Group: 800mg Ibuprofen (Intrafen Flk, Gen drug, Turkey) in 150 ml normal saline given as a slow intravenous infusion over 5 minutes.
* Drug packs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the paracetamol or Ibuprofen medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered as a infusion over 5 minutes.
* Randomization was achieved by using computer software to generate random numbers.
* One researcher blinded to patient allocation observed the whole procedure and recorded the Low Back Pain scores.
* Patients in both groups received two types of medication in a similar manner (for example, 150 ml normal saline given as a slow intravenous infusion over 5 minutes), thus ensuring double blinding.
* Low Back Pain scores were recorded at 0, 15, and 30 min on a VAS of 1 to 10
* Rescue medication is given within 30 minutes after study drug administration if the patients say yes that question "Do you need any additional analgesic requirement".
* All other medications required during the study also were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with complaints of low back pain to the emergency services ,
* Patients whose complaints have started in the last week,
* Younger than 21 years old,
* older than 80 years old,

Exclusion Criteria:

* Pretreatment linear 100-mm visual analog scale (VAS) pain score less than 40 mm,
* Patients who have drop foot, paralysis and other neurological symptoms in physical examination.
* Patients with blood pressure less than 90mmHg in the arrival of emergency services.
* Patients with malignancy, cauda equina syndrome, ankylosing spondylitis, rheumatoid arthritis or inflammatory arthritis contain any of the disease in his/her CV.
* Patients with any history of chronic pain syndrome.
* Patients who receive pain killers, antidepressants, anticonvulsants, muscle relaxants, steroids within 6 hours before the ED visit,
* Patients have a history of active peptic ulcer disease,
* Patients who have signs of peritoneal irritation,
* Patients had a fever (>37.9)
* Allergy or previous adverse reaction to the studied drugs(Ibuprofen, Paracetamol), received agents to inhibit the secretion of acid (PPIs or histamine-2 receptor antagonists), antispasmodics, or nonsteroidal anti-inflammatory drugs
* were pregnant or breast-feeding,
* inability to comprehend the VAS evaluation,
* or refused to participate in the study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of Low Back Pain on the Visual Analog Scale | Low Back Pain scores will be recorded at 0, 15, and 30 min on a VAS of 1 to 10

SECONDARY OUTCOMES:
Adverse events | 30th minutes after the study drug administered
  30th minutes after the study drug administered

IPD SHARING:
Plan to Share IPD: Undecided